CLINICAL TRIAL: NCT01365949
Title: INI-1 Deletions in Ewing Sarcoma
Brief Title: Biomarker in Tissue Samples From Patients With Ewing Sarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEWS11B1; COG-AEWS11B1 (Other: Children's Oncology Group); NCI-2011-02857 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AEWS11B1 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Sarcoma
Keywords: Ewing sarcoma/peripheral primitive neuroectodermal tumor (PNET)
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: microarray analysis
Genetic: protein analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in tissue samples from patients with Ewing sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the frequency of INI-1 protein loss in Ewing Sarcoma.

OUTLINE: Previously collected tissue samples are analyzed for INI-1 protein loss by IHC and tissue microarray.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Ewing sarcoma
* Prepared tissue microarray with Ewing sarcoma samples available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of Ewing sarcoma.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-05; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Frequency of INI1 protein loss in Ewing Sarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D. Schiffman, MD, Principal Investigator — University of Utah